CLINICAL TRIAL: NCT02192489
Title: A Phase 2A, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Sequential, Dose-Ascending Study Of CC-220 In Subjects With Chronic Cutaneous Sarcoidosis
Brief Title: A Phase 2 Study With CC-220 in Skin Sarcoidosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-220-SAR-001; 2014-001065-27 (EudraCT Number)
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Sarcoidosis
Keywords: Chronic Cutaneous Sarcoidosis; Cutaneous Sarcoidosis; Skin Sarcoidosis; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — iberdomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CC-220 0.3mg (Experimental): CC-220 0.3 mg capsules by mouth (PO) daily for 12 weeks
  Interventions: Drug: CC-220 0.3 mg Daily
- CC-220 0.6mg (Experimental): CC-220 0.6mg capsules by PO daily for 12 weeks
  Interventions: Drug: CC-220 0.6mg Daily
- Placebo (Placebo Comparator): Identically matching placebo PO daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-220 0.3 mg Daily
  Arms: CC-220 0.3mg
Drug: CC-220 0.6mg Daily
  Arms: CC-220 0.6mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of oral CC-220 in adult subjects with chronic cutaneous sarcoidosis.

DETAILED DESCRIPTION:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, sequential, dose-ascending, safety and tolerability study in subjects with chronic cutaneous sarcoidosis.

Two dose cohorts of CC-220 (Cohort 1: 0.3 mg by mouth (PO) every day (QD) or matching placebo and Cohort 2: 0.6 mg PO QD or matching placebo) will be evaluated using a sequential, dose-ascending design

ELIGIBILITY:
Inclusion Criteria:

Males or females aged ≥ 18 years at the time of consent.

* Have chronic cutaneous sacrcoidosis (CCS) prior to consent
* Have active cutaneous sarcoidosis lesion(s) at screening
* Forced vital capacity of ≥ 45% of predicted normal value at screening.
* Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min.
* Females of childbearing potential must have negative pregnancy tests prior to starting study therapy and agree to either commit to true abstinence or use effective contraception.
* Male subjects must practice true abstinence or agree to use a condom even if he has undergone a successful vasectomy

Exclusion Criteria:

* Positive tuberculosis test at screening.
* History of inadequately treated tuberculosis
* History of Human Immunodeficiency Virus (HIV) and/or Common Variable Immunodeficiency Disease.
* History of alcohol or drug abuse
* History or current peripheral neuropathy
* Current uveitis or any other clinically significant ophthalmological finding
* Currently require therapy for precapillary pulmonary hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11-01 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 12 weeks
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health.

SECONDARY OUTCOMES:
Improvement in modified Sarcoidosis Activity and Severity Index | Week 4, 8 and 12
  Proportion of subjects who achieve a ≥ 1-point change in the index lesion as measured by the cutaneous sarcoidosis outcome instrument (modified Sarcoidosis Activity and Severity Index) as compared to baseline
Improvement in lesion induration | Week 12
  Change from baseline in lesion induration via dermascope compared to Week 12
Improvement in sarcoidosis disease markers | Weeks 4, 8, 12
  Change from baseline in sarcoidosis disease markers: serum angiotensin converting enzyme (ACE), Immunoglobulin G (IgG) levels, 25-hydroxy vitamin D (25-OH-vit D), and 1,25-dihydroxy vitamin D (1,25-vit D) as compared to Weeks 4, 8 and 12.
Pharmacokinetics- Maximum Plasma Concentration (Cmax) of CC-220 After Single and Multiple Doses | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  Maximum observed plasma concentration after a single dose on Day 1 or multiple doses on Day 29).
Pharmacokinetics - Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Time Point After Single and Multiple Doses (AUC 0-t) | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  Area under the plasma concentration time-curve from time 0 to the last quantifiable concentration at time t following a single dose (day 1) and multiple doses (Day 29) determined using the trapezoidal method (non-compartmental analysis).
Pharmacokinetics - Area Under the Plasma Concentration-time Curve From Time Zero to Infinity After Single and Multiple Doses (AUC0-inf) | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  The area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) for CC-220 after a single dose on day 1 and multiple doses on Day 29, calculated by the linear trapezoidal rule and extrapolated to infinity.
Pharmacokinetics - Terminal Phase Half-life (t1/2) After Single and Multiple Doses | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  Terminal phase elimination half-life (t1/2) after a single dose on day 1 and multiple doses on Day 29
Pharmacokinetics - Apparent Volume of Distribution (Vz/f) After Single and Multiple Doses | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  Apparent volume of distribution after a single dose on day 1 and multiple doses on Day 29, based on the terminal phase after a orally administration
Pharmacokinetics - Apparent Total Clearance of CC-220 (CL/F) After Single and Multiple Doses | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  The apparent total clearance after a single dose on Day 1 and multiple doses Day 29, calculated as Dose/AUC0-inf
Pharmacokinetics - Time to Maximum Plasma Concentration (Tmax) After Single and Multiple Doses | Day 1 and Day 29 at predose, 1, 2, 3, 4, 6, 8, and 24 hours post-dose
  The time to first maximum observed plasma concentration of CC-220 after a single dose (Day 1) or multiple doses (Day 29).

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, MD, PhD, Study Director — Celgene Corporation